CLINICAL TRIAL: NCT06660862
Title: DAROSTEP: Evaluating Step Counts as a Biomarker and Its Relationship on Treatment Outcomes in Vulnerable Patients With Metastatic Hormone-Sensitive Prostate Cancer on Darolutamide and Androgen Deprivation Therapy
Brief Title: Evaluating Treatment Outcomes Using Darolutamide and Androgen Deprivation Therapy in Patients With Metastatic Hormone-Sensitive Prostate Cancer.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0691
Record Dates: First submitted 2024-09-11; First posted 2024-10-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — darolutamide; Hormones; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Darolutamide and physical activity correlation (Experimental): To understand how darolutamide plus hormone therapy affects physical activity, we would like to specifically monitor the step count of men receiving these medications.
  Interventions: Drug: Darolutamide; Drug: Physician choice Androgen Deprivation (Hormone) Therapy

INTERVENTIONS:
Drug: Darolutamide — How darolutamide and hormone therapy affects the step count of older men who have prostate cancer
Drug: Physician choice Androgen Deprivation (Hormone) Therapy — How step count/physical activity affects certain quality of life changes these men experience such as differences in pain, mood, function, memory and fatigue

SUMMARY:
This prospective clinical trial aims to investigate the impact of darolutamide in combination with standard-of-care androgen deprivation on physical activity, specifically step count, and its correlation with important markers of safety in vulnerable adults who screen positive by a brief geriatric assessment (GA) and metastatic hormone-sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged ≥18 years.
* Patients must exhibit an ECOG performance status of ≤3.
* Patients must screen positive for frailty by having ONE of the following:

  1. Katz Activities of Daily Living (ADL) Assessment Score 3 or 4 out of 533.
  2. 4-Instrumental activities of daily living (4-IADL) assessment score 2 or 3 out of 4 34.
  3. A Grade 3 event on the Cumulative Illness Score Rating-Geriatrics (CISR-G) questionnaire35 (excluding prostate cancer.)
  4. Body mass index (BMI) ≤21 kg/m² and/or >10% weight loss in the last 6 months
* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.

  a) Patients without histologic evidence of prostate cancer are eligible if have documented metastatic disease and PSA>50ng/dL
* Patients must have at least one metastatic bone and/or soft tissue/visceral lesion documented in the following manners within 42 days prior randomization:

  1. Metastatic disease to the bone (in any distribution) visible on 99Tc-MDP bone scintigraphy or PSMA-PET on either pre-ADT scans or baseline scans AND/ OR
  2. Lymph node metastases of any size or distribution (PSMA-PET positive or 1.5cm in short access to support metastatic prostate cancer diagnosis).
  3. Visceral metastases of any size or distribution. If a participant has a history of visceral metastases at any time prior to randomization, he should be coded as having visceral metastases at baseline (i.e., patients with visceral metastases prior to ADT that disappear at baseline will be counted as having visceral metastases and would therefore have high volume disease for stratification purposes).
* Patients must have adequate organ function:

  1. Bone marrow reserve ANC ≥1.5 x 109/L Platelets ≥100 x 109/L, Hemoglobin ≥8 g/dL [transfusion of PRBC or PLT for eligibility purposes only will not be allowed]
  2. Hepatic: Total bilirubin ≤2 x the institutional upper limit of normal (ULN), for patients with known Gilbert's Syndrome ≤3 x ULN is permitted. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3.0 x ULN OR ≤5.0 x ULN for patients with liver metastases
* Testosterone ≥100 mg/dL
* Albumin ≥2.5 g/dL
* Patients eligible for this study must be either:

  1. Completely untreated (treatment-naïve) for metastatic prostate cancer.
  2. Minimally treated, which includes:

     1. Use of LHRH agonists/antagonists or bilateral orchiectomy, with or without a first-generation antiandrogen (e.g., bicalutamide, flutamide), for up to 45 days prior to joining the study.
     2. Any first-generation antiandrogen must be stopped before beginning the study treatment or within 45 days of starting these treatments, whichever is earlier.
* Patients must consent and concurrently accrue to the IRONMAN registry study (NCT03151629)
* If patient is a sexually active male and/or his female partner is of childbearing potential, patient must agree to use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) from screening through 3 months after the last dose of study drugs.

Exclusion Criteria:

* Patients who have previously received any ADT or ARSI within 12 months of metastatic diagnosis are not eligible.

  a) Patients who received ADT and/or ARSI for locally advanced disease or in an adjuvant or salvage setting are eligible, provided this treatment was not within 12 months before their metastatic diagnosis.
* Uncontrolled intercurrent illness includes ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, bed-bound status, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

  a. Patients with eGFR <15 or on dialysis are excluded
* Participants with known small-cell carcinoma of the prostate or known brain metastasis.
* Participants with limb defects precluding accelerometer wear.
* Any prior systemic anti-prostate cancer therapy (with the exception of the drugs listed on inclusion criteria), including chemotherapy, Poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitors, immunotherapy or biological therapy (including monoclonal antibodies).
* Concurrent cytotoxicity chemotherapy, immunotherapy, radioligand therapy, PARP inhibitor, biological therapy or investigational therapy
* Previous treatment with any of the following within 6 months of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation or other PSMA-targeted radioligand therapy is not allowed
* Ongoing participation in any other treatment clinical trial. Concurrent accrual to non-treatment trials such as biomarker or registry trials is allowed.
* Use of other investigational drugs within 30 days prior to day of randomization
* Known hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes
* Diagnosed with other malignancies that require active treatment or may interfere with disease assessment.
* Active clinically significant cardiac disease defined as any of the following:

  1. NYHA class 3/4 congestive heart failure within 6 months prior to ICF signature unless treated with improvement and echocardiogram or MUGA demonstrates EF > 45% with improvement in symptoms to class < 3.
  2. History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants in the study such as: Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, complete left bundle branch block, high-grade atrioventicular (AV) block (e.g., bifascicular block, Mobitz type II and third degree AV block)
  3. Cardiac or cardiac repolarization abnormality, including any of the following: History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to ICF signature
* Inability to complete the study imaging procedures due to any reason (e.g., severe claustrophobia, inability to lie still for the entire imaging time, any condition that precludes raised arms position)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Investigating the impact of darolutamide in combination with ADT on step count | 6 months
  To investigate the impact darolutamide in combination with ADT on the physical activity (digitally collected step count) of vulnerable adults with metastatic hormone-sensitive prostate cancer over a 6-month treatment period.

SECONDARY OUTCOMES:
Step count and the Global Health Score | 12 months
  To examine the relationship between step count and the Global Health Score from the EORTC QLQ-C30.
Physical Function | 3, 6, 9, and 12 months.
  To examine the relationship between step count and the Physical Function subscale from the EORTC QLQ-C30.
Fatigue subscale | 3, 6, 9, and 12 months.
  To examine the relationship between step count and the Fatigue subscale from the EORTC QLQ-C30.
Pain Severity | 3, 6, 9, and 12 months.
  To examine the relationship between step count and Pain Severity from the Brief Pain Inventory (BPI).
Occurrence of serious adverse events | 12 months
  To relate step count to the occurrence of serious adverse events over 12 months of treatment with darolutamide + ADT.
Digitally collected step count | 12 months
  To investigate the impact of darolutamide with ADT on digitally collected step count at 12 months of treatment.
Geriatric assessment parameters | 12 months
  To investigate the impact of darolutamide with ADT on geriatric assessment parameters by G-CODE over a 12-month interval.
Safety of darolutamide with ADT | 12 months
  To characterize the safety of darolutamide with ADT in vulnerable adults captured through assessment of adverse events by CTCAE v5.0.
Mobility ability | 3, 6, 9, and 12 months
  To investigate the effect of darolutamide with ADT on mobility, measured by the Timed Up and Go (TUG) test.
Grip strength ability | 3, 6, 9, and 12 months
  To investigate the effect of darolutamide with ADT on grip strength, measured using a dynamometer.
Lower-body strength ability | 3, 6, 9, and 12 months
  To investigate the effect of darolutamide with ADT on lower-body strength, measured using the Chair Stand Test.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, Principal Investigator — University of Chicago Medicine Comprehensive Cancer Center
Locations (1):
- o University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States